CLINICAL TRIAL: NCT00626717
Title: Riboflavin Mediated Corneal Crosslinking for Stabilizing Progression of Keratoconus
Acronym: CCL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Collaborators: Peschke Meditrade, GmbH (Industry)
Responsible Party: Principal Investigator, D Dr. Philip Maier, PD Dr. med., University Hospital Freiburg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FR-03-CCL
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Keratoconus
Keywords: Keratoconus; Cross linking; Riboflavin
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Procedure: Riboflavin/UVA crosslinking
- 2 (Sham Comparator)
  Interventions: Procedure: Sham treatment

INTERVENTIONS:
Procedure: Riboflavin/UVA crosslinking — Removal of epithelium. Riboflavin eye drops. UVA exposure.
  Arms: 1
Procedure: Sham treatment — Fluorescein eye drops. Exposure with blue light
  Arms: 2

SUMMARY:
Background: Corneal cross linking is a procedure that induces collagen cross linking of the corneal stroma due to release of reactive oxygen radicals upon activation of topically applied riboflavine A by UVA exposure. This procedure might be capable of reducing keratocouns progression.

Purpose: Although there are no randomised controlled trials on the effectiveness of corneal cross linking for the treatment of keratoconus it gains more and more importance in the general clinical setting. Therefore, the investigators started such randomised, placebo controlled, double blinded, multicenter trial to find out if this treatment is as effective as it promises to be.

Methods: Randomised, placebo controlled, double blinded, multicenter trial.

ELIGIBILITY:
Inclusion Criteria:

* Only early Keratoconus (Contact lens fitting)
* Progression of Ametropia.
* Corneal thickness > 450µm

Exclusion Criteria:

* Further ophthalmic diseases
* History of ocular surgery
* Pregnancy, brest feeding
* Allergy against Riboflavin
* End stage Keratoconus

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Keratoconus progression | 3 years
Endothelial cell loss | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Philip Maier, MD, Principal Investigator — University Eye Hospital, Freiburg
Locations (1):
- University Eye Hospital Freiburg, Freiburg im Breisgau, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Lang SJ, Messmer EM, Geerling G, Mackert MJ, Brunner T, Dollak S, Kutchoukov B, Bohringer D, Reinhard T, Maier P. Prospective, randomized, double-blind trial to investigate the efficacy and safety of corneal cross-linking to halt the progression of keratoconus. BMC Ophthalmol. 2015 Jul 21;15:78. doi: 10.1186/s12886-015-0070-7. PMID 26194634